CLINICAL TRIAL: NCT04807712
Title: National Surveillance of Pediatric Pertussis in Ambulatory Settings
Brief Title: Pediatric Pertussis in Ambulatory Settings
Acronym: ACTIVCOQ
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: GlaxoSmithKline (Industry); Sanofi (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ACT0606
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Pertussis/Whooping Cough; Children, Only; Ambulatory
Keywords: Pertussis; surveillance; pertussis acellular vaccine
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional study

SUMMARY:
Since 2002, Whooping cough surveillance in pediatric private practice has been set up in France. The results of the first years, 2002-2006, have confirmed the effectiveness of the Pertussis whole-cell (Pw) vaccine and in particular the duration of protection of 9/10 years. After evaluating cases in children vaccinated with Pw vaccines, the study aims today to analyze cases in children vaccinated with Pertussis acellular (Pa) vaccines used since 2002/2003 and to assess, on an outpatient basis, the impact of new vaccine recommendations in France (in 2013, introduction of a 2 + 1 schedule - 8 weeks, 4 months and a 11-month recall - and a 6-year recall, and in 2014, update in the recommendations of exams to be prescribed based on the child's age and vaccination status).

DETAILED DESCRIPTION:
The whooping cough surveillance objectives are :

* to follow the duration of protection of the Ca vaccines in the context of modifications of the vaccine recommendations
* to describe the clinical characteristics of a population vaccinated with several boosters
* to adapt complementary examinations for diagnostic purposes (culture, PCR, serology) according to the evolution of scientific knowledge
* to monitor B. parapertussis infections
* to train laboratories with nasopharyngeal aspiration
* to monitor the evolution of the bacterial species All children aged 0-18 years, in whom the diagnosis of pertussis is mentioned and for which a biological check-up is requested, are included, except asymptomatic children with confirmed family case.

In case of suspected pertussis, real-time PCR and / or culture and / or (rarely) serology is / are still prescribed to the patient and / or his entourage.

Selected Pediatricians from the ACTIV group and the AFPA working in an outpatient clinic, located in different places in France, are participating in this network since 2001. The clinical evolution and the results of the examinations are transcribed on a case report form. The data are collected, firstly, during the visit where the diagnosis of whooping cough is suspected and a biological assessment requested (patient's medical history, clinical data, vaccination status and dates, as well as the search for a contaminated/contaminator) and secondly during the follow-up visit (results of the biological check-up and diagnosis, antibiotics potentially prescribed, and supplement data of the entourage, except in case of diagnosis of pertussis not retained).

All evaluations made by the pediatricians are regularly reviewed during meetings, and final diagnoses used are:

* biological pertussis
* epidemiological pertussis
* not evaluable
* lost of follow up
* no whooping cough

ELIGIBILITY:
Inclusion Criteria:

* All children under 18 years old with a pertussis diagnosis is suspected and a biological exam is requested

Exclusion Criteria:

* children without symptoms with a household confirmed case
* cases for which the pertussis diagnosis was not suspected by the pediatrician

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children under 18 years with suspected pertussis diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 898 (Estimated)
Dates: Start 2001-05-30 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Duration of pertussis vaccines protection | at inclusion
  Evaluate the duration of protection of the Ca vaccines

SECONDARY OUTCOMES:
Clinical characteristics of pertussis | at inclusion
  Describe the clinical characteristics of a population vaccinated

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Guiso, Study Director — Institut Pasteur
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Whooping cough surveillance in France in pediatric private practice in 2006-2015 — https://pubmed.ncbi.nlm.nih.gov/28974408/
- See also: Pertussis surveillance in private pediatric practices, France, 2002-2006 — https://pubmed.ncbi.nlm.nih.gov/18598649/
- See also: Guidelines for diagnosis of whooping cough — https://pubmed.ncbi.nlm.nih.gov/14550985/